CLINICAL TRIAL: NCT05341206
Title: Evaluation the Effects of Herbal Gargle for Chemoradiotherapy-induced Oral Mucositis of Head & Neck Cancer, a Pilot Study.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202101017A3
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Neoplasms; Chemoradiotherapy; Stomatitis and Ulceration
Keywords: Medicine, Chinese Traditional; Head and Neck Neoplasms; Chemoradiotherapy; Stomatitis and Ulceration
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Ulcer | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The treatment group receive Herbal gargle and control group receive normal saline.
Masking Description: The color of Herbal gargle is yellowish while normal saline is transparent. Therefore, the study belongs to open label trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group receive Herbal gargle 150ml and are instructed to hold the gargle in the mouth for 30s and then expectorate it twice a day, 5 days a week for 8 weeks.
  Interventions: Drug: Herbal gargle
- Control group (Sham Comparator): The control group receive Normal saline 150ml and are instructed to hold the normal saline in the mouth for 30s and then expectorate it twice a day, 5 days a week for 8 weeks.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Herbal gargle — The treatment group receive Herbal gargle 150ml and are instructed to hold the gargle in the mouth for 30s and then expectorate it twice a day, 5 days a week for 8 weeks.
  Arms: Treatment group
Other: Normal saline — The control group receive Normal saline 150ml and are instructed to hold the normal saline in the mouth for 30s and then expectorate it twice a day, 5 days a week for 8 weeks.
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate the effects of Herbal gargle on chemoradiotherapy-induced stomatitis in head & neck cancer patients.

DETAILED DESCRIPTION:
Head and neck cancer accounts for about 5% of all cancers worldwide with the age-standardized incidence rate (ASIR) of HNC increased by 5.4% per year among males and 3.1% among females in Taiwan. Concurrent chemoradiotherapy (CCRT) is the most common management to treat head and neck cancer. However, CCRT may cause much side effects such as oral mucositis, radiation dermatitis, xerostomia, or infection, which influence food intake, disturb nutritional status and interrupt the course of treatment. Traditional Chinese Medicine (TCM) has been applied to treat cancer side effects for many years. Herbal gargle is composed of TCM herbals used for oral mucositis induced by chemoradiotherapy among head and neck cancer. The aim of the trial is to evaluate the effectiveness of Herbal gargle. The participants divide into two groups, treatment group and control group. The treatment group receive Herbal gargle 150ml and are instructed to hold the gargle in the mouth for 30s and then expectorate it twice a day, 5 days a week for 8 weeks. The control group receive normal saline 150ml for oral mucositis. The subjective questionnaires of EORTC QLQ-C30, EORTC QLQ-H&N35 are assessed twice a week, CTCAE for grading of oral mucositis is assessed once a week, VAS is assessed everyday for 8 weeks. Besides, change of opioid dosage, body weight are also recorded. The CRP is assessed before and every week for 8 weeks and the albumin and bacteria culture are assessed before and post-treatment of 4th week and 8th week. The baseline difference of treatment and control group will be analyzed by using independent t-test and the difference of evaluation scores and blood tests between pre-treatment and post-treatment will be analyzed using multivariate logistic regression analysis. A value of P < 0.05 will be regarded as statistically significant for the above statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Willing to join the trial project and sign the informed consent form.
* Age more than 20 years-old.
* Pathology proved to be head and neck cancers.
* Head and neck cancer patients under radiotherapy or concurrent chemoradiotherapy.
* Expected life expectancy more than 3 months.
* Subjects with clear consciousness and can be assessed cooperatively.
* Subjects are suitable to use Herbal gargle evaluated by Traditional Chinese medicine physicians.

Exclusion Criteria:

* Subjects can not sing the informed consent form.
* Systemic infection.
* Heart, liver and kidney insufficiency
* Allergy history of Traditional Chinese medicine
* Unclear conscious to use Herbal gargle.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of CTCAE 4.0 | change from baseline and every week for 8 weeks.
  CTCAE is used to describe the severity of oral mucositis for patients receiving cancer therapy.

SECONDARY OUTCOMES:
Change of EORTC QLQ-C30 | change from baseline at 4 weeks and 8 weeks post treatment.
  European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire score, EORTC QLQ-C30, is used to measure cancer patients' physical, psychological and social functions.
Change of EORTC QLQ-H&N35 | change from baseline at 4 weeks and 8 weeks post treatment.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-head & neck, EORTC QLQ-H&N35, is used for assessing the health-related quality of life for head-and-neck cancer patients.
Change of VAS of pain of oral mucositis | change from baseline and everyday for 8 weeks.
  Visual Analogue Scale, VAS, is used to to measure the intensity of pain of oral mucositis.
Change of body weight | change from baseline and every week for 8 weeks.
  The oral mucositis caused by chemoradiotherapy will influence food intake. Monitor body weight provides objective evaluation of nutrition status.
Change of opioid use | change from baseline and every week for 8 weeks.
  Opioid analgesics is often prescribed for alleviating pain from oral mucositis. Monitor opioid use provides other evaluation for severity of pain and wound healing.
Change of albumin | change from baseline at 4 weeks and 8 weeks post treatment.
  Albumin has been used as maker of nutrition status.
Change of CRP | change from baseline and every week for 8 weeks.
  C-reactive protein is used to monitor severity of oral mucositis.
Change of common aerobic culture | change from baseline and every week for 8 weeks.
  Aerobic culture is used to monitor the change of bacteria flora before and after Herbal gargle treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Keelung, Taiwan, Taiwan